CLINICAL TRIAL: NCT04112368
Title: Cyclical Neuroactive Steroid Changes, Arousal, and Proximal Suicide Risk: An Experimental Approach
Acronym: CLEAR-3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Tory Anne Eisenlohr-Moul, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2019-0624
Record Dates: First submitted 2019-09-25; First posted 2019-10-02 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation | interventions — Estradiol; Progesterone; Sugars

STUDY DESIGN:
Intervention Model Description: Crossover 2-Condition Placebo-Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Identical placebos provided by the University of Illinois at Chicago investigational drug service.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transdermal Estradiol + Oral Micronized Progesterone (Experimental): 0.1 mg/24hr transdermal estradiol patch applied weekly and 100 mg oral micronized progesterone taken twice daily by mouth, for 14 days starting 7 days after a positive urine luteinizing hormone (LH) test.
  Interventions: Drug: Estradiol Transdermal Patch 0.1 mg/24 hrs; Drug: Oral Micronized Progesterone 200mg; Drug: Inactive Clear Patch; Drug: Placebo capsule
- Placebo Patch + Placebo Pills (Experimental): Placebo patch (selected to match transdermal estradiol patch) applied weekly and placebo pills (blinded to match oral micronized progesterone) taken twice daily by mouth, for 14 days starting 7 days after a positive urine luteinizing hormone (LH) test.
  Interventions: Drug: Estradiol Transdermal Patch 0.1 mg/24 hrs; Drug: Oral Micronized Progesterone 200mg; Drug: Inactive Clear Patch; Drug: Placebo capsule

INTERVENTIONS:
Drug: Estradiol Transdermal Patch 0.1 mg/24 hrs — Estradiol transdermal patch delivering 0.1 mg/24 hour administered by affixing to skin for 14 days starting on day 7 after ovulation
  Other Names: Climara
Drug: Oral Micronized Progesterone 200mg — 100 mg oral micronized progesterone taken orally twice daily for 14 days starting day 7 after ovulation (200mg total per day)
  Other Names: Prometrium
Drug: Inactive Clear Patch — Matching placebo patch administered by affixing to skin for 14 days starting on day 7 after ovulation
  Other Names: Placebo transdermal patch
Drug: Placebo capsule — Matching placebo capsules administered twice daily for 14 days starting day 7 after ovulation
  Other Names: Sugar pill

SUMMARY:
Female suicide attempts occur more often in the weeks before and after menses onset, and have been linked to ovarian hormone withdrawal. The proposed project will use a two-week intervention to stabilize hormones in females with recent suicidal thoughts; this paradigm is a safe way to learn how cyclical changes in hormones and their metabolites influence short-term risk of suicide. The data acquired will contribute to our understanding of the biology of acute suicide risk and advance efforts to develop safe and effective treatments that eliminate predictable monthly worsening of suicide risk in reproductive-age females.

DETAILED DESCRIPTION:
Suicide is the second leading cause of death among women of reproductive age, and female suicide attempts occur most frequently around menses (perimenstrually), when estradiol (E2) and progesterone (P4) fall rapidly. A recent prospective study demonstrated that suicidal ideation (SI) and attempts peak perimenstrually in natural cycles, and that this perimenstrual worsening of SI can be prevented by administering stabilizing doses of E2+P4 (relative to placebo). Therefore, while E2+P4 withdrawal is a viable model of proximal suicide risk in females with SI, mechanisms are unclear. GABAergic neuroactive steroid metabolites of ovarian hormones (e.g., allopregnanolone), exert potent sedative and antidepressant effects; we hypothesize that acute perimenstrual withdrawal from these hormone metabolites may increase suicide risk by increasing hyperarousal and hopelessness. The long-term objectives of this research are to (1) use the menstrual cycle as a model to probe the proximal mechanisms of suicide, and (2) develop long-term treatments that eliminate hormonal contributions to suicide. The objective of the current work is to use a crossover placebo-controlled trial of E2+P4 stabilization (vs. natural E2+P4 withdrawal under placebo) in the perimenstrual weeks to probe behavioral (hopelessness, hyperarousal) and molecular/genetic (neuroactive steroid levels, mRNA expression for enzymes critical for synthesizing neuroactive steroids) mediators of perimenstrual suicide risk. Design: In this mechanistic trial, 90 female outpatients with past-month SI will complete two counterbalanced conditions: (1) two weeks of placebo during natural perimenstrual E2+P4 withdrawal, and (2) two weeks of perimenstrual E2+P4 stabilization (.1mg/day transdermal estradiol + 200mg/day oral micronized progesterone) to prevent withdrawal. Five labs per condition will capture changes in gas chromatography mass spectrometry (GC-MS) quantified neuroactive steroids, messenger ribonucleic acid (mRNA) expression for enzymes critical for synthesizing neuroactive steroids, and physiological arousal. Our app (BiAffect) will collect ecological momentary assessments (EMA; 4x/day) of behavioral constructs and SI, and will passively track arousal via movement and typing speed instability. Specific Aims. Aim 1 is to evaluate hyperarousal and hopelessness as interacting mechanisms by which perimenstrual E2+P4 withdrawal (vs. experimental E2+P4 stabilization) increases proximal suicide risk. Aim 2 is to evaluate neuroactive steroid withdrawal as a mechanism by which perimenstrual E2+P4 withdrawal (vs. stabilization) increases proximal suicide risk. If appropriate, a multilevel path model will test a path in which E2+P4 withdrawal (vs. stabilization) causes neuroactive steroid withdrawal, which increases in hopelessness and hyperarousal, which in turn increases proximal suicide risk. Relevance. By conducting a mechanistic experiment to probe the mediators of a known cause of proximal suicide risk, the proposed research responds to public calls from the National Institute of Mental Health (NIMH)-sponsored Suicide Research Prioritization Agenda to identify modifiable causes of proximal suicide risk.

ELIGIBILITY:
Inclusion Criteria:

* Ability to adhere to medication regimen
* Speaks English
* Assigned female at birth with intact ovaries
* Premenopausal
* Normal menstrual cycles between 25-35 days
* Under current care of an outpatient mental health provider with visits occurring at least once every 3 months.
* At least 1 year postpartum.
* Willing to use a barrier method of birth control during the study.
* Normal weight (BMI between 18-29)
* Must report at least some recent suicidal ideation (in the past month) at the time of recruitment.
* Must be categorized as having acceptably low imminent risk for suicidal crisis/attempt by a licensed clinical psychologist utilizing evidence-based clinical and research guidelines for imminent suicide risk management.

Exclusion Criteria:

* Must not be pregnant, breastfeeding, or trying to become pregnant.
* Must not be taking any form of exogenous hormones or hormonal intrauterine device, and must have ended previous use of hormonal preparations at least one month prior to the study.
* Must not have a personal history of any chronic medical condition, including but not limited to metabolic or autoimmune disease, epilepsy, endometriosis, cancer, diabetes, cardiovascular, gastrointestinal, hepatic, renal, or pulmonary disease, and no personal or first degree family history of thromboembolic events.
* Any current cigarette smoking is exclusionary.
* Must not report a history of clinical diagnosis or treatment for postpartum depression or premenstrual dysphoric disorder (Note: Premenstrual Dysphoric - - - Disorder diagnosis must have been made based on prospective daily ratings).
* Must not report any history of manic episode, any history of psychotic symptoms, or current substance use disorder.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Since the study is focused on the menstrual cycle, the study includes only those assigned female sex at birth
Enrollment: 124 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tory A Eisenlohr-Moul, Ph.D, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Neuropsychiatric Institute, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Condition, Then Inactive Condition: Beginning 7 days after ovulation, active treatment begins 7 days after ovulation with an estradiol transdermal patch (0.1 mg/24 hrs) applied to the skin weekly (spanning 14 days of treatment) along with (active) 100 mg oral micronized progesterone capsules taken twice daily by mouth for 14 days. A 1-month washout is observed. Then, beginning 7 days after ovulation, inactive placebo capsules will be taken twice daily by mouth along with the application of inactive clear patches applied to the skin weekly for 14 days.
- Inactive Condition, Then Active Condition: Beginning 7 days after ovulation, inactive placebo capsules will be taken twice daily by mouth along with the application of inactive clear patches applied to the skin weekly for 14 days. After completing a 1-month washout, active treatment begins 7 days after ovulation with an (active) estradiol transdermal patch applied to the skin weekly (spanning 14 days of treatment) along with (active) 100 mg oral micronized progesterone capsules taken twice daily by mouth for 14 days.
Period: Overall Study
Arm/Group | Active Condition, Then Inactive Condition | Inactive Condition, Then Active Condition
Started | 61 | 63
Completed | 41 | 44
Not Completed | 20 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Condition, Then Inactive Condition | Inactive Condition, Then Active Condition | Total
Number analyzed (Participants) | 61 | 63 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 63 | 124
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 63 | 124
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 21 | 37
  Not Hispanic or Latino | 44 | 42 | 86
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 34 | 25 | 59
  More than one race | 10 | 8 | 18
  Unknown or Not Reported | 4 | 16 | 20
Region of Enrollment [Number; unit: Participants]
  United States | 61 | 63 | 124

OUTCOME MEASURES:

1. Primary Outcome: Perimenstrual Change in Daily Adult Suicidal Ideation Questionnaire (ASIQ) Scores
Description: The Adult Suicidal Ideation Questionnaire (ASIQ) is a 25-item self-report questionnaire assessing suicidality. Each day, individuals rate each of 25 items on a scale from 1 (Not at All) to 6 (Extreme). Mean scores are computed, providing a single number for each day that represents the participant's mean suicidal ideation (1 to 6), with higher daily values representing more severe suicidal ideation.
  Perimenstrual change scores are calculated for each person in each condition as the mean of scores in the perimenstrual phase (days +12 to +17 following a positive luteinizing hormone surge in urine on day=0) minus the mean in the midluteal phase (days +0 to +5). Therefore, positive values represent a perimenstrual increase in suicidal ideation, and negative values represent a perimenstrual decrease.
Time Frame: Mean daily rating in the perimenstrual phase (days +12 to +17 following a positive luteinizing hormone surge in urine on day=0) minus the mean daily rating in the midluteal phase (days +0 to +5)
Measure: Mean (Standard Error); unit: Mean Score Change
Groups:
- Placebo Patch + Pills: Placebo patch manufactured to mimic transdermal estradiol applied weekly and placebo pills manufactured to mimic oral micronized progesterone taken twice daily by mouth, for 14 days starting 7 days after a positive urine luteinizing hormone (LH) test.
Arm/Group | Placebo Patch + Pills | Transdermal Estradiol + Oral Micronized Progesterone
Number analyzed (Participants) | 85 | 85
Mean Score Change | .178 (.08) | -.051 (.05)
Statistical Analysis 1: Comparison: Placebo Patch + Pills vs Transdermal Estradiol + Oral Micronized Progesterone; Fixed interaction effect of treatment (0=Placebo, 1=E2+P4) by cycle phase (0=Lower-Risk Baseline, 1=Higher-Risk Perimenstrual Phase) predicting SI severity in a multilevel model (with daily observations nested within conditions nested within participants over time); Test type: Superiority; p < .001, Mixed Models Analysis; This is the p-value for the Treatment X Cycle Phase Interaction. Kenward-Roger Method was utilized for degrees of freedom; Slope = -.02, 95% CI 2-sided [-.02 to -.02]

2. Primary Outcome: Perimenstrual Change in Daily Columbia Suicide Severity Rating Scale (C-SSRS) Screening Interview Planning Item Scores
Description: The Columbia Suicide Severity Rating Scale is an interview designed to assess various aspects of suicide risk. In the present study, this questionnaire is administered daily via phone interview as part of a risk screening process. Here, we utilize a single dichotomous outcome from a single item representing suicidal planning from the C-SSRS interview: "Today, have you thought about how or when you might kill yourself?". Each day, individuals chose either "Yes" (coded as 1) or "No" (coded as 0).
  Perimenstrual change scores are calculated for each person in each condition as the mean of scores in the perimenstrual phase (days +12 to +17 following a positive luteinizing hormone surge in urine on day=0) minus the mean in the midluteal phase (days +0 to +5). Therefore, positive values represent a perimenstrual increase in suicidal planning, and negative values represent a perimenstrual decrease.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: Mean Score Change
Arm/Group | Transdermal Estradiol + Oral Micronized Progesterone | Placebo Patch + Placebo Pills
Number analyzed (Participants) | 85 | 85
Mean Score Change | -.04 (.02) | .021 (.008)
Statistical Analysis 1: Comparison: Transdermal Estradiol + Oral Micronized Progesterone vs Placebo Patch + Placebo Pills; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .026, Mixed Models Analysis; Slope = .19, 95% CI 2-sided [.04 to .82]

3. Secondary Outcome: Perimenstrual Change in Daily Beck Hopelessness Scale (BHS) Short Form Scores
Description: Hopelessness is assessed with a daily Beck Hopelessness Scale (short form), a 10-item self-report measure with true-false items that assess hopelessness and the extent of positive and negative beliefs about the future. Summed scores range from 0 to 10. Scores provide a measure of the severity of self-reported hopelessness, with higher scores representing greater hopelessness.
  Perimenstrual change scores are calculated for each person in each condition as the mean of scores in the perimenstrual phase (days +12 to +17 following a positive luteinizing hormone surge in urine on day=0) minus the mean in the midluteal phase (days +0 to +5). Therefore, positive values represent a perimenstrual increase in hopelessness, and negative values represent a perimenstrual decrease.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: Mean Score Change
Arm/Group | Transdermal Estradiol + Oral Micronized Progesterone | Placebo Patch + Placebo Pills
Number analyzed (Participants) | 85 | 85
Mean Score Change | -.004 (.003) | .25 (.06)
Statistical Analysis 1: Comparison: Transdermal Estradiol + Oral Micronized Progesterone vs Placebo Patch + Placebo Pills; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .052, Mixed Models Analysis; Slope = -.09, 95% CI 2-sided [-.18 to .00]

4. Secondary Outcome: Perimenstrual Change in Daily Brief Agitation Measure (BAM) Scores
Description: Agitation is assessed with a daily Brief Agitation Measure (BAM), a 3-item self-report measure in which participants rate their symptoms of agitation ranging from 0 (Strongly Disagree) to 6 (Strongly Agree). Mean daily scores (ranging from 0 to 6) provide a measure of the severity of self-reported agitation, with higher scores representing greater agitation.
  Perimenstrual change scores are calculated for each person in each condition as the mean of scores in the perimenstrual phase (days +12 to +17 following a positive luteinizing hormone surge in urine on day=0) minus the mean in the midluteal phase (days +0 to +5). Therefore, positive values represent a perimenstrual increase in agitation, and negative values represent a perimenstrual decrease.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: Mean Score Change
Arm/Group | Transdermal Estradiol + Oral Micronized Progesterone | Placebo Patch + Placebo Pills
Number analyzed (Participants) | 85 | 85
Mean Score Change | -.066 (.015) | .005 (.003)

ADVERSE EVENTS:
Time Frame: Daily using a standardized checklist during the 14 days of treatment in each condition.
Arm/Group | Transdermal Estradiol + Oral Micronized Progesterone | Placebo Patch + Placebo Pills
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/106
Other Adverse Events (participants affected / at risk) | 77/111 | 64/106
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdermal Estradiol + Oral Micronized Progesterone (N=111) | Placebo Patch + Placebo Pills (N=106)
Skin Irritation (Skin and subcutaneous tissue disorders) | 35 (35) | 12 (12)
Breast Discomfort (Reproductive system and breast disorders) | 24 (24) | 11 (11)
Joint Pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 8 (8)
Perceived Negative Emotional Changes (Psychiatric disorders) | 15 (15) | 19 (19)
Nausea (Gastrointestinal disorders) | 16 (16) | 13 (13)
Dizziness (General disorders) | 9 (9) | 3 (3)
Vision Changes (Eye disorders) | 5 (5) | 2 (2)
Chest Discomfort (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Headache (General disorders) | 17 (17) | 10 (10)
Venipuncture Bruising (Skin and subcutaneous tissue disorders) | 7 (7) | 11 (11)
Perceived Change in Menses (Reproductive system and breast disorders) | 11 (11) | 1 (1)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT04112368/Prot_001.pdf
  • Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT04112368/SAP_000.pdf